CLINICAL TRIAL: NCT01292070
Title: A Dose-Escalating Phase 0 Study to Evaluate the Safety and Local Cutaneous Reactivity of Intradermal Human Fcγ1-Fel d1 Fusion Protein (GFD) in Cat-allergic Healthy Volunteers
Brief Title: Safety Evaluation of an Experimental Treatment, Intradermal Human Fcγ1-Fel d1 Fusion Protein (GFD), for Cat Allergy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Futility
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Tunitas Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN048AD
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-01

CONDITIONS: Cat Allergy
Keywords: Fel d 1 protein, Felis domesticus; Injections, Intradermal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control-Experimental arm (Experimental): Each subject will serve as their own control with the left arm receiving the control protein (Histamine prick, intradermal diluent and intradermal CAT) and right arm receiving the experimental protein (GFD).
  Interventions: Biological: Intradermal Human Fcγ1-Fel d1 fusion protein; Biological: Positive Control - standardized cat hair allergenic extract (CAT); Biological: Positive Control - Histamine Prick; Biological: Negative Control - Intradermal Diluent

INTERVENTIONS:
Biological: Intradermal Human Fcγ1-Fel d1 fusion protein — Part A: 7 sequential 10-fold dose increments from 0.001 BAU/mL to 1,000 BAU/mL; An 8th dose of 10,000 BAU/mL might be given only if the 10 BAU/mL of CAT is the dose that elicits a bump or hive of >= to 10mm.
  Part B: 5 sequential 10-fold dose increments from 0.1 BAU/mL to 1,000 BAU/mL; An 6th dose of 10,000 BAU/mL might be given only if the 10 BAU/mL of CAT is the dose that elicits a bump or hive of >= to 10mm.
Biological: Positive Control - standardized cat hair allergenic extract (CAT) — 4 sequential 10-fold injections starting from 0.01 BAU/mL to 10 BAU/mL
Biological: Positive Control - Histamine Prick — 1.0 mg/mL
  Other Names: Histatrol GLY
Biological: Negative Control - Intradermal Diluent — Saline, Albumin with Phenol (HSA) sterile diluent

SUMMARY:
The purpose of this trial is to show that Intradermal Human Fcγ1-Fel d1 fusion protein (GFD) is able to block the skin reaction to cat allergen in cat allergic subjects compared to the skin reaction to cat allergen alone. This research project is also testing the safety and tolerability of this new, experimental treatment, compared to the current treatment of cat allergen alone.

DETAILED DESCRIPTION:
Researchers are conducting a research study of a new protein developed to treat sensitivity to cat allergens. Cat allergy in humans is an allergic reaction to one or more of the five known allergens produced by cats. The most common of these is the protein Fel d 1.

This study will test Intradermal Human Fcγ1-Fel d1 fusion protein (GFD), a new protein that, based on animal data, has been developed to block the allergic effects of cat. If this drug works the way they think it does, it may become a treatment for cat allergy that is faster than the currently available treatments and with fewer side effects. This protein contains the molecule from the cat, that causes the allergic reaction, attached to a section of a particular antibody (protein involved in immunity) called Fcγ1 that acts like a break. The fusion of the two proteins is predicted to interrupt the flow of cellular reactions which lead to the allergic response.

This will be the first time GFD is administered to humans. The study will be conducted in two parts. The subjects in part A will be administered intradermal standardized cat hair allergenic extract (CAT) and GFD sequentially in 10-fold increasing doses every 20 minutes. If Part A demonstrates the safety of GFD,subject in part B will begin by following the same treatment as part A followed by a rechallenge of the sites with CAT at 4 hours after the first dose of GFD. Each subject will be evaluated 3 times (screening, dosing, and telephone follow-up 2 days post dosing) and will return on Day 28 for blood draw.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic reactivity to cats as expressed by allergic rhinitis
* Radioallergosorbent test (RAST test) for cat-specific IgE with RAST rating of 2 (0.70-3.49 KU/L IgE) documented within the past year or at screening
* Standardized cat hair allergenic extract (CAT), 10,000 BAL/mL (ALK-Abello) elicits a wheal 5 mm or greater than the diluent control (Saline Albumin with Phenol [HSA], ALK-Abello) with surrounding erythema on testing using a standardized epicutaneous delivery device (Stallergenes Prick Lancet, 1 mm tip)
* Histamine (Histatrol 1mg/mL, ALK-Abello) reactivity of 5 mm or greater reactivity than the diluent control with surrounding erythema on epicutaneous testing using a standardized epicutaneous delivery device
* Able and willing to discontinue any anti-histamine use for 5 days prior to entry into protocol and throughout the protocol participation
* Baseline spirometry (FEV1, FVC FEF25-75) with FEV1 >=80% predicted and other values within the normal range
* Ability to give written informed consent

Exclusion Criteria:

* Diluent control (Saline Albumin with Phenol [HSA], ALK-Abello) elicits wheal >= 3 mm on epicutaneous testing using a standardized epicutaneous delivery device
* Pregnant females as determined by a positive serum or urine hCG test
* Lactating females
* Ever having received allergen immunotherapy (e.g., -subcutaneous allergen [SCIT] or -sublingual [SLIT])
* Systemic steroids in the past 3 months
* Severe systemic reactivity on exposure to cats (e.g., laryngeal or angioedema, fainting, pallor, bradycardia, hypotension, bronchospasm, asthma, or generalized urticaria)
* A clinical history of asthma
* Underlying heart, liver, kidney lung, or other medical condition (acute infections, immune diseases, current substance abuse) such that the person would be at a clearly increased risk for a poor outcome should a generalized allergic reaction occur
* Use of systemic beta-blocking or ACE-inhibiting agents within the past 3 weeks
* Use of tri-cyclic antidepressants within the past 3 weeks
* Subjects receiving therapy with any agents known or likely to interact with adrenaline (e.g., beta blockers, ACE-Inhibitors, tri-cyclic antidepressants, or other)
* Current use or use of omalizumab (Xolair) within past 6 months
* Subjects with any extensive skin disorder (atopic dermatitis) that would make skin testing or proper interpretation impractical
* Mental impairment, limiting the ability to comply with study requirements
* Participation in a clinical trial and receipt of an investigational product within 30 days, 5 half-lives or twice the duration of the biochemical effect of the investigational product (whichever is longer) prior to dosing in the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Saxon, MD, PhD, Study Chair — University of California, Los Angeles
Locations (1):
- Alfred Hospital and Monash University, Melbourne, Victoria, Australia

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/Pages/default.aspx
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One center in Australia recruited four participants with a history of allergic reactivity to cats as expressed by allergic rhinitis and who had reactivity to standardized cat hair allergenic extract
Groups:
- Control (CAT) - Experimental (GFD): Each participant served as their own control: the left arm received the control protein (histamine prick, intradermal diluent and intradermal standardized cat hair allergenic extract (CAT)) and right arm received the experimental protein (human Fcgamma1-Fel d1 (cat allergen) fusion protein (GFD)) administered intradermally (ID). The control arm received CAT at 0.02 milliliters (mL) of 0.01 bioequivalent allergy units (BAU)/mL to 10 BAU/mL (sequentially in 10-fold increments, stopping if dose produced a wheal ≥ 10 millimeters (mm)). The experimental arm received GFD at 0.001 BAU/mL (1/10th the dose of Fel d1 in the lowest dose of CAT) administered at 0.02 mL. Dosing continued sequentially in 10-fold increments until either a wheal of ≥ 10 mm or the maximum dose was reached (maximum of 7 dose increments).
Period: Overall Study
Arm/Group | Control (CAT) - Experimental (GFD)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Arm/Group | Control (CAT) - Experimental (GFD)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (2.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  Australia | 4

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Doses of GFD and CAT Required to Elicit a Cutaneous Reaction Demonstrated by a Wheal Greater Than or Equal to 10 mm With Surrounding Erythema
Description: Difference in the doses of human Fcgamma1-Fel d1 (cat allergen) fusion protein (GFD) and standardized cat hair allergenic extract (CAT) required to elicit a wheal ≥ 10 mm with surrounding erythema.
Time Frame: up to 3 hours after the last injection of GFD
Population: The experimental protein (human Fcgamma1-Fel d1 fusion protein (GFD)) and the control protein (standardized cat hair allergenic extract (CAT)) elicited comparable reactivity in the first four participants dosed; thus, the trial was discontinued for futility and the primary endpoint was not evaluated
Arm/Group | Control (CAT) - Experimental (GFD)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Start of study through Day 28
Description: Adverse events severities were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (published May 28, 2009 and updated to 4.02 on September 15, 2009). Wheal, erythema, and pruritus at site of administration were expected outcomes and thus were not reported as adverse events
Arm/Group | Control (CAT) - Experimental (GFD)
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (CAT) - Experimental (GFD) (N=4)
Rhinitis (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The experimental protein (human Fcgamma1-Fel d1 fusion protein) & control protein (standardized cat hair allergenic extract) elicited comparable reactivity in the first four participants dosed and consequently the trial was discontinued for futility

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No